CLINICAL TRIAL: NCT04285411
Title: Results of the SpO2 and Pulse Rate Accuracy Comparison of VitalDetect™ to Arterial Blood CO-Oximetry and Reference ECG
Brief Title: Vital USA SpO2 Accuracy Comparison to Arterial Blood CO-Oximetry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vital USA, Inc. (Industry)
Collaborators: Clinimark, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: PR 2019-353
Record Dates: First submitted 2020-02-23; First posted 2020-02-26 (Actual); Results first posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Arterial Disease

STUDY DESIGN:
Intervention Model Description: Testing was conducted under normal office environment conditions. The VitalDetect™ pulse oximetry was placed on the right index finger of all subjects to evaluate the SpO2 and pulse rate accuracy performance during steady state non-motion conditions. A Control Pulse Oximetry system was also placed on the subject to evaluate the stability of the draws and the real time oxygen saturation status. The subject was in a reclined position and connected to a breathing circuit, for administering medical grade oxygen and nitrogen. The gas flow delivery was adjusted for subject comfort. Arterial blood samples were drawn during simultaneous data collection from the control pulse oximeter and the test oximeters. The blood was immediately analyzed by Reference CO-Oximetry providing functional SpO2 for the basis of the SpO2 accuracy comparison. The pulse rate for the VitalDetect™ was compared to Reference ECG Heart Rate collected during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- ARMS SpO2 70-100% (Experimental): Comparison to Reference CO-Oximetry
  Interventions: Device: Accuracy of the VitalDetect™ pulse oximetry system

INTERVENTIONS:
Device: Accuracy of the VitalDetect™ pulse oximetry system — The purpose of this study was to validate the SpO2 accuracy of the VitalDetect™ pulse oximetry system during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-Oximetry. It was expected that the Accuracy Root Mean Square (ARMS) performance of the oximetry system would meet the required specification of ARMS of 3.0% or less.

SUMMARY:
Clinical Investigation Plan: Vital USA SpO2 Accuracy Comparison to Arterial Blood CO-Oximetry Study ID# PR 2019-353, Version: Rev 1, Date: 15 Oct 2019 Study Dates: November 4-5, 2019

DETAILED DESCRIPTION:
An SpO2 accuracy comparison was conducted as part of the final validation of the VitalDetect™ pulse oximetry system. The study was conducted in accordance to Code of Federal Regulations (CFR) for Non-Significant Risk (NSR) investigational studies, following International Standards Organization (ISO) 14155:2011 as appropriate and the pulse oximetry guidelines of ISO 80601-2-61:2017 applicable sections, and Pulse Oximeters - Premarket Notifications Submissions [510(k)s] Guidance For Industry and Food and Drug Administration Staff (issued: March 4, 2013).

The purpose of this study was to validate the SpO2 accuracy of the VitalDetect™ pulse oximetry system during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-Oximetry. It was expected that the Accuracy Root Mean Square (ARMS) performance of the oximetry system would meet the required specification of ARMS of 3.0% or less.

A secondary goal was to evaluate the pulse rate performance simultaneously collected over the SpO2 range covered. The Pulse Rate Accuracy Root Mean Square (Arms) performance of the VitalDetect™ pulse oximetry system, were expected to meet a specification of 3 bpm.

ELIGIBILITY:
Inclusion Criteria

1. 10-15 Adults with a minimum of 3 males and a minimum of 3 females, with the balance made up of either
2. Subject must have the ability to understand and provide written informed consent
3. Subject is 18 to 50 years of age
4. Subject must be willing and able to comply with study procedures and duration
5. Subject is a non-smoker or who has not smoked within 2 days prior to the study

Exclusion Criteria

1. Subject is considered as being morbidly obese (defined as BMI >39.5).
2. Compromised circulation, injury, or physical malformation of fingers, wrist, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the particular sites utilized.)
3. Female subjects that are actively trying to get pregnant or are pregnant (confirmed by positive urine pregnancy test unless the subject is known to be not of child-bearing potential).
4. Smoker Subjects who have refrained will be screened for COPD levels >3% as assessed with a Radical 7 (Rainbow)
5. Subjects with known respiratory conditions such as: (self-reported):

   1. uncontrolled / severe asthma,
   2. flu,
   3. pneumonia / bronchitis,
   4. shortness of breath / respiratory distress,
   5. unresolved respiratory or lung surgery with continued indications of health issues,
   6. emphysema, COPD, lung disease.
6. Subjects with known heart or cardiovascular conditions such as: (self-reported, except for blood pressure and ECG review)

   1. hypertension: systolic >140mmHg, Diastolic >90mmHg on 3 consecutive readings (reviewed during health screen).
   2. have had cardiovascular surgery
   3. Chest pain (angina)
   4. heart rhythms other than a normal sinus rhythm or with respiratory sinus arrhythmia (reviewed during health screen)
   5. previous heart attack
   6. blocked artery
   7. unexplained shortness of breath
   8. congestive heart failure (CHF)
   9. history of stroke
   10. transient ischemic attack
   11. carotid artery disease
   12. myocardial ischemia
   13. myocardial infarction
   14. cardiomyopathy
7. Self-reported health conditions as identified in the Health Assessment Form (self-reported)

   1. diabetes,
   2. uncontrolled thyroid disease,
   3. kidney disease / chronic renal impairment,
   4. history of seizures (except childhood febrile seizures),
   5. epilepsy,
   6. history of unexplained syncope,
   7. recent history of frequent migraine headaches,
   8. recent symptomatic head injury (within the last 2 months)
   9. cancer / chemotherapy
8. Subjects with known clotting disorders (self-reported)

Ages: 18 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Ruiz, MD, Principal Investigator — Avista Adventist Hospital
Locations (1):
- Clinimark Laboratory Services, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Following Institutional Review Board (IRB) approval Title: "Vital USA SpO2 Accuracy Comparison to Arterial Blood CO-Oximetry", Clinimark Study ID# PR 2019-353, eleven healthy adult volunteer subjects were screened and enrolled into the study. One subject was withdrawn due to poor device placement and time sync with the control oximeter.
Period: Overall Study
Arm/Group | ARMS SpO2 70-100%
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 10 Healthy volunteer subjects of five (5) males and five (5) females ages 19-38 years, weight 105-228 lbs, height 63-75 inches, and BMI 18 - 34.7. Two (2) Black/ African Americans, one (1) Asian, and seven (7) White. Nine (9) Non-Hispanic/Non-Latino and one (1) Hispanic / Latino.
Arm/Group | ARMS SpO2 70-100%
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.9 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Skin tone [Count of Participants; unit: Participants]
  Light Skin Tone | 4
  Medium Light Skin tone | 2
  Medium Skin Tone | 1
  Dark Skin Tone | 3
Weight [Mean (Standard Deviation); unit: Lbs] | 161.0 (41.4)
Height [Mean (Standard Deviation); unit: inches] | 68.4 (4.2)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.0 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Evaluate SpO2 Accuracy Per Standards for Pulse Oximetry.
Description: This study was a comparative, single-center, non-randomized study conducted to evaluate the SpO2 accuracy per standards and guidelines identified above for SpO2 accuracy for pulse oximetry equipment over the range of 70-100% SaO2 under non-motion conditions. Arterial blood sampling measured by functional SaO2 CO-Oximetry, was used as the basis for comparison. As a secondary goal, the pulse rate accuracy was compared to ECG Heart Rate realized over the range throughout the hypoxia procedure. Testing was conducted under normal office environment conditions.
Time Frame: 90 Seconds
Population: Five (5) males, five (5) females (age: 19-38yrs, weight: 105-228 lbs, height: 63-75", BMI: 18.0-34.7). Race ethnicity, two (2) Black / African-Americans, one (1) Asian, seven (7) White. Nine (9) Non-Hispanic / Non-Latino, one (1) of Hispanic /Latino. Skin pigmentation ranged from light to dark meeting the requirement of at least 2 darkly pigmented
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | ARMS SpO2 70-100%
Number analyzed (Participants) | 10
percent | 3.1 (0.6)

2. Secondary Outcome: The Pulse Rate Accuracy Compared to ECG Heart Rate.
Description: The pulse rate accuracy was compared to ECG Heart Rate as recorded by the S5 Multi-parameter monitor. Passing criteria was an ARMS of 3 bpm or better based measurements observed during the pulse oximetry evaluation.
Time Frame: 90 Seconds
Population: Five (5) males, five (5) females (age: 19-38yrs, weight: 105-228 lbs, height: 63-75", BMI: 18.0-34.7). Race / ethnicity, two (2) Black / African-Americans, one (1) Asian, seven (7) White. Nine (9) Non-Hispanic / Non-Latino, one (1) Hispanic /Latino. Skin pigmentation / tones met requirement of at least 2 darkly pigmented or 15 % of the subject pool
Measure: Mean (Standard Deviation); unit: percent
Groups:
- ARMS SpO2 70-100%: Compared to ECG Heart Rate.
Arm/Group | ARMS SpO2 70-100%
Number analyzed (Participants) | 10
percent | 2.7 (06)

ADVERSE EVENTS:
Time Frame: up to 15 days after the completion of the study
Description: All subjects completed the study without incidence.
Groups:
- ARMS SpO2 70-100%: Comparison to Reference CO-Oximetry
  Accuracy of the VitalDetect™ pulse oximetry system: The purpose of this study was to validate the SpO2 accuracy of the VitalDetect™ pulse oximetry system during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-Oximetry. It was expected that the Accuracy Root Mean Square (ARMS) performance of the oximetry system would meet the required specification of ARMS of 3.0% or less.
  No Adverse events reported
Arm/Group | ARMS SpO2 70-100%
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT04285411/Prot_SAP_000.pdf